CLINICAL TRIAL: NCT04114409
Title: The Prevalence of Type D Personality in OSAS and the CPAP Therapy Compliance and Cardiovascular Complications in Moderate to Severe OSAS With Type D Personality.
Brief Title: Type D Personality and the Compliance for CPAP Therapy and Cardiovascular Complications in OSA.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Sonia De Weerdt, medical physician, Universitair Ziekenhuis Brussel
Other Study IDs: Slaaplabo protocol doc
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-08

CONDITIONS: Academic Underachievement Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: OSAS and type D personality
- 2: OSAS without type D personality

SUMMARY:
Type D personality is characterized by negative affectivity and social inhibition and is assessed with the DS-14 questionnaire. This type of personality was initially described in patients with coronary heart disease and associated with poor prognosis and diminished quality of life. Whereas the prevalence of type D personality in patients with coronary heart disease is between 27% and 31%, the prevalence in the general population is between 13% and 24%. The prevalence of type D personality in OSA (Obstructive Sleep Apnea Syndrome) was only investigated in patients with a moderate or severe OSA (Apnea-hypopnea index > 15/hour) already on standard clinical treatment with CPAP (Continuous Positive Airway Pressure). The overall prevalence of type D personality in OSA is still unknown. Furthermore, OSA is frequently associated with cardiovascular disease. No studies were performed on the impact of type D personality and cardiovascular complications in OSA.

Until now, only a few studies were performed to investigate type D personality in OSA patients treated with CPAP therapy. One retrospective study showed that OSA patients with type D personality experienced more side effects of CPAP treatment and were less compliant to therapy. In a more recent prospective study, the influence of type D personality on CPAP compliance could not be confirmed. No information is available about the frequency of visits and the time spent by these patients to remediate CPAP side effects. There is also no data about the discontinuation rate of CPAP treatment in this population of patients. It is possible that a specific follow up of those patients is needed to enhance CPAP compliance.

After a while, CPAP therapy can have an influence on mood and behavior. Therefore, it is possible that CPAP therapy can alter the patient's answers to the DS-14 questionnaire. This could explain the different outcome of the retrospective and prospective studies mentioned above. No studies were performed to test the reliability and validate the DS-14 questionnaire in OSA patients.

Consequently, the aim of the present study is to evaluate more extensively the importance of type D personality traits in OSA patients.

DETAILED DESCRIPTION:
Objective of the study

1. To determine the overall prevalence of type D personality in untreated OSA ( Obstructive sleep apnea) patients and their subtypes; mild, moderate, severe and REM (rapid eye movement) OSA.

   Full polysomnography and questionnaires:ESS, PSQI, DS-14, SF-36, ISI, FAS, HADS, BFI-2, CIS will be used to answer this question.

   A multistage tracking for gender and type D personality was done. In general population, there are twice as much men than women suffering from OSA. This means that the investigator need to recruit 41% (√ 2 ≈ 1.41%) more men than women. In the general population, the prevalence of type D personality is 25%.

   To answer this question, the investigator also assume that there will be 50 % mild, 25% moderate and 25% severe OSA.

   Chi- squared test:

   With a power of 0.9: 97 type D patients are needed with a total of 400 patients to be recruited.
2. To establish the reliability and validity of the DS-14 questionnaire to diagnose type D personality in OSA patients.

   Full polysomnography and questionnaires:ESS, PSQI, DS-14, SF-36, ISI, FAS, HADS, BFI-2, CIS will be used. the DS-14 questionnaire will be filled out one month later.

   An interclass correlation analysis with kappa ≈ 0.8 will give a good correlation between the two scores. First, a pilot study will be done on a small sample of patients. In function of these results, a sample calculation required to have a significant result will be done. In an earlier study, 135 patients with type D personality were studied to assess the reproducibility of the DS-14 questionnaire.
3. To investigate the impact of type D personality on CPAP ( continuous positive airway pressure) treatment in OSA patients, especially on compliance for CPAP, on the CPAP discontinuation rate and on the frequency and time spent to remediate side effects of CPAP treatment.

   Full polysomnography and questionnaires:ESS, PSQI, DS-14, SF-36, ISI, FAS, HADS, BFI-2, CIS will be used. The DS-14 questionnaire will be filled out one month later.Titration polysomnography 2 months later and questionnaires: ESS, PSQI, DS-14, SF-36, ISI, FAS, HADS, CIS.Consultation 3 month later for control compliance and questionnaires: DS-14, SF-36, HADS, FAS, CIS, EES, PSQI.Polyclinic visit 1 year later for control compliance and questionnaires: DS-14, SF-36, HADS, FAS, CIS, EES, PSQI.Monitoring time and frequency of free consultation for resolving any side effects of the CPAP treatment.

   Additionally, the investigator assume that there is a 25% chance (midrange) to discontinue CPAP treatment and 70% (midrange) compliance. Compliance will be normalized to a percentage scale by dividing by the expected hours of sleep (for the power analysis, we take 7 hours expected sleep). A hypothetical difference of 1 hour will therefore represent 14.29% (=1/7).

   For the t-tests:

   Standard deviation: based on a 95% interval for CPAP [4h-9h], the investigator divide this interval of 5 h by 4 (4 sigma's for 95%). Followed by a normalization (1/7), one sigma gives 17.86%. With a power of 0.9 and α= 0.01 (Bonferonni correction), 128 patients will be needed for an unbalanced design of both groups in a ratio of 75% versus 25%.

   For the Fisher Exact- test:

   General OSA population Expected in type D Good compliance 70% (between 60 & 80%) 56% ( 70% minus 14%) Poor compliance 30% 44%

   With a power of 0.9: in total 580 patients are needed. (580 patients of which 25% type D: Feasible since about 500 new OSA patients are diagnosed and treated a year at the UZ Brussels)
4. To determine the influence of type D personality on cardiovascular complications in OSA.

Baseline polysomnography: two groups: OSA with type D and without type D and questionnaires: ESS, PSQI, DS-14, SF-36, ISI, FAS, HADS, BFI-2, CIS. Search medical files for cardiovascular morbidity in both groups Additionally, the investigator assume that there is a 25% chance (midrange) to discontinue CPAP treatment and 70% (midrange) compliance. Compliance will be normalized to a percentage scale by dividing by the expected hours of sleep (for the power analysis, we take 7 hours expected sleep). A hypothetical difference of 1 hour will therefore represent 14.29% (=1/7).

For the t-tests:

Standard deviation: based on a 95% interval for CPAP [4h-9h], the investigator divide this interval of 5 h by 4 (4 sigma's for 95%). Followed by a normalization (1/7), one sigma gives 17.86%. With a power of 0.9 and α= 0.01 (Bonferonni correction), 128 patients will be needed for an unbalanced design of both groups in a ratio of 75% versus 25%.

For the Fisher Exact- test:

General OSA population Expected in type D Good compliance 70% (between 60 & 80%) 56% ( 70% minus 14%) Poor compliance 30% 44%

With a power of 0.9: in total 580 patients are needed. (580 patients of which 25% type D: Feasible since about 500 new OSA patients are diagnosed and treated a year at the UZ Brussels)

Procedures To determine the overall prevalence of type D personality in untreated OSA patients and their subtypes, all patients admitted to the sleep laboratory for a polysomnography will be asked to participate to this study. An informed consent will be signed and patients will complete a number of questionnaires. In the current practice of the sleep laboratory, the Epworth sleepiness scale, the Stanford sleepiness scale, the Pittsburgh sleep quality index, the Insomnia severity scale, the DS-14 questionnaire, the SF-36 questionnaire, the FAS, HADS, BFI-2 and CIS are filled out by each patient.

All patients who test positive for OSA (AHI > 5/hour) and positive for type D personality (DS-14: SI>10 and NA>10) will be asked to complete these questionnaires once more 1 month later. This is necessary to evaluate the test-retest reliability/stability of the DS-14 questionnaire in OSA. To evaluate the validity of this questionnaire in OSA, correlation patterns with the BFI-2 and the HADS will be investigated.

For all patients diagnosed with moderate OSA in which treatment with CPAP is indicated, the questionnaires will be repeated during their second polysomnography (standard of care), 3 months after the second polysomnography (standard of care) and 1 year after this last visit (standard of care). The second polysomnography is needed to estimate the therapeutic pressure and to meet the criteria for the OSA convention. The time necessary for treatment education (time to explain function of CPAP), frequency of visits and time necessary to deal with complications, treatment compliance (hours of use CPAP device), treatment discontinuation will be monitored. The group with OSA and type D personality will be compared with the OSA group without type D personality.

A search for cardiovascular events in the electronic medical file of all OSA patients with and without type D personality will be carried out.

The above mentioned procedures will all be carried out in the sleep laboratory of the UZ Brussel, Laarbeeklaan 101, 1090 Jette.

ELIGIBILITY:
Inclusion Criteria:

* All patients with an OSA (AHI (Apnea-hypopnea index) >5/hour) and type D personality (DS- 14 score: SI (social inhibition) >10 and NA (negative affectivity) >10)
* Age > 18 years

Exclusion Criteria:

* - Age < 18 years
* AHI< 5/hour
* All patients incapable to understand the study or to sign the informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients attending the sleeplaboratory
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
The overall prevalence of type D personality in untreated OSA ( Obstructive sleep apnea) patients and their subtypes; mild, moderate, severe and REM (rapid eye movement) OSA. | 4 years
  The prevalence of type D personality in the different types of OSA wil be statistically calculated after scoring the DS-14 questionnaire as wel as other questionnaires, ESS, PSQI, SF-36, ISI, FAS, HADS, BFI-2, CIS. These questionaires will be filled out by the population patients refered to the sleeplaboratory for a full polysomnography.
The reliability and validity of the DS-14 questionnaire to diagnose type D personality in OSA patients. | 4 years
  The DS-14 questionnaire, filled out at baseline polysomnography will be repeated 1 month later and the scores will be compared by an interclass correlation analysis. This is necessary for the reliability. For the validity of the questionnaire, a correlation between the BFI-2 will be necessary
the impact of type D personality on CPAP ( continuous positive airway pressure) treatment in OSA patients on compliance for CPAP, CPAP discontinuation rate and frequency and time spent to remediate side effects of CPAP treatment. | 4years
  The questionnaires, ESS, PSQI, DS-14, SF-36, ISI, FAS, HADS, BFI-2, CIS, filled out at baseline polysomnography will be repeated during the titration night ( night necessary to evaluate pressure and for the convention OSA). During the different required visits , some of these questionnaires will be repeated ( see above). The scores of these questionnaires will be compared during CPAP therapy. The compliance of therapy ( registrated automatically by the CPAP devise) will be compared between two groups, OSA + type D and OSA without type D. The time spend for education of the use of the cpap, the time necessary to solve complication of therapy and the frequency of visits to the sleeplaboratory of the patients in both groups will be recorded and compared. Allso the discontinuation of cpap therapy will be compared in both groups.
To determine the influence of type D personality on cardiovascular complications in OSA. | 4years
  In both groups (OSA+ type D and OSA without type D) a search in the medical file for cardiovascular events in the history will be done by recording arythmias, hypertension, cerebrovascular accident. The results will be compared between the two groups